CLINICAL TRIAL: NCT05882786
Title: Comparing the Efficacy of Corticosteroid Injection and Tendon Dry Needling for Subacromial Impingement Syndrome: A Randomized Clinical Trial
Brief Title: Corticosteroid Injection Versus Tendon Dry Needling for Subacromial Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ImpDn1
Record Dates: First submitted 2023-05-07; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome; Shoulder Impingement; Subacromial Impingement Syndrome; Subacromial Impingement
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome | interventions — Adrenal Cortex Hormones; Dry Needling

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The corticosteroid (Triamcinolone Acetonide) injection group (Active Comparator): Participants in this group will receive a single subacromial injection of 40mg triamcinolone acetonide.
  Interventions: Procedure: Corticosteroid injection
- Tendon dry needling group (Active Comparator): Participants in this group will receive a total of 3 sessions of dry needling treatment to the supraspinatus, infraspinatus, and subscapularis muscle tendons.
  Interventions: Procedure: Dry Needling

INTERVENTIONS:
Procedure: Corticosteroid injection — Subacromial injection of 40mg triamcinolone acetonide.
  Arms: The corticosteroid (Triamcinolone Acetonide) injection group
Procedure: Dry Needling — Dry needling treatment to the supraspinatus, infraspinatus, and subscapularis muscles tendons.
  Arms: Tendon dry needling group

SUMMARY:
This randomized clinical trial aims to compare the efficacy of corticosteroid injection and tendon dry needling for the treatment of subacromial impingement syndrome.

DETAILED DESCRIPTION:
This randomized clinical trial will compare the efficacy of corticosteroid injection and tendon dry needling for the treatment of subacromial impingement syndrome.Participants will be randomized to receive either a corticosteroid injection or tendon dry needling treatment. The corticosteroid injection group will receive a single subacromial injection of 40mg triamcinolone acetonide under ultrasound guidance. The tendon dry needling group will receive a total of 3 sessions of dry needling treatment to the supraspinatus, infraspinatus, and subscapularis muscle tendons. Patients will be assessed before treatment, after treatment, after three weeks and after three months with visual analog scale, Shoulder Pain and Disability Index (SPADI) and shoulder range of motion measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years old
* Diagnosis of subacromial impingement syndrome, confirmed by clinical examination and imaging (such as X-ray or MRI)
* Moderate to severe shoulder pain, with a score of at least 4 on a 0-10 visual analog scale (VAS) for pain
* Willingness to comply with the study protocol and attend all study visits and assessments
* Ability to provide informed consent to participate in the study.

Exclusion Criteria:

* Contraindications to corticosteroid injection or dry needling, such as local infection, bleeding disorders, or allergy to the injectate or needle
* Previous shoulder surgery on the affected shoulder
* Other active shoulder conditions, such as rotator cuff tear or adhesive capsulitis, that may confound the study results
* Systemic conditions, such as rheumatoid arthritis or osteoarthritis, that may affect the shoulder joint and its function
* History of shoulder dislocation or instability
* Pregnancy or breastfeeding
* Current use of systemic corticosteroids or immunosuppressive drugs
* Injection to shoulder area in the past six months.
* Inability to complete the study assessments or follow the study protocol, such as due to cognitive impairment or language barrier.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale for Pain | First day, after three weeks, after three months
  A Visual Analog Scale (VAS) for pain is a commonly used tool to measure the intensity of pain experienced by a patient. It typically consists of a horizontal or vertical line, typically 10 centimeters long, with endpoints labeled as "no pain" and "worst possible pain." The patient is asked to mark on the line the point that best represents the intensity of their pain, with the distance from the "no pain" end of the line to the patient's mark representing the pain score.
Change in The Shoulder Pain and Disability Index (SPADI) | First day, after three weeks, after three months
  The Shoulder Pain and Disability Index (SPADI) is a validated patient-reported outcome measure that is commonly used to assess pain and functional disability related to shoulder disorders. The SPADI consists of 13 items that assess pain and disability in two domains: 1) pain and 2) disability. The pain domain consists of five items that assess the intensity and frequency of shoulder pain, while the disability domain consists of eight items that assess the impact of shoulder pain on daily activities such as sleeping, dressing, and carrying objects.
Change in Range Of Motion (ROM) Measurements | First day, after three weeks, after three months
  ROM of the shoulder joint is typically assessed using a goniometer, a device that measures joint angles. The goniometer is used to measure the degree of movement in different directions, including flexion, extension, abduction, adduction, internal rotation, and external rotation. The measurements obtained from the goniometer can then be used to determine the improvement or deterioration in ROM over time, which can be an indicator of treatment efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon reasonable request by the corresponding author.
Supporting Information: Study Protocol, CSR
Time Frame: 1 month.
Access Criteria: Individual participant data will be shared upon reasonable request by the corresponding author.